CLINICAL TRIAL: NCT00614406
Title: The Effects of a Prostaglandin Inhibitor on Ovulation and the Menstrual Cycle.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Alison Edelman, MD, MPH, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: OHSU FAMPLAN 3854
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Ovulation (Follicular Rupture Yes/no); Menstrual Cycles (Total Length, Bleeding Days); Gonadotropin and Ovarian Hormone Levels (FSH, LH, E2, P)
Keywords: Celebrex; prostaglandin inhibitor; ovulation; menstrual cycles
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Celebrex
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Celebrex — One 400mg tablet daily.
  Arms: 1
Drug: Placebo — One tablet daily.
  Arms: 2

SUMMARY:
The investigators propose to test the hypothesis that the use of a prostaglandin inhibitor will result in premature luteolysis (ovulation failure) in women.

DETAILED DESCRIPTION:
Currently available methods of emergency contraception (EC) only work during a very narrow time period prior to the hormonal trigger for ovulation or the release of an egg. Women having unprotected sex outside this window receive no benefits from this emergency therapy. Prostaglandins are critical before, during, and after ovulation, thus their inhibition may cause an EC effect that works over a longer time period. We wanted to determine if celecoxib might work as an EC with a wider window of action.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Normal menstrual periods (24-35 days)
* Good general health
* Willing to use a non-hormonal form of contraception for the entire study (Acceptable forms of contraception include condoms, spermicide, sexual contact with a sterilized partner, subject is surgically sterile, same-sex partner, Copper IUD and abstinence)
* Willing and able to return to clinic for bi-weekly blood tests

Exclusion Criteria:

* Pregnant or breast feeding
* Polycystic ovarian disease
* Gastrointestinal conditions (i.e.gastric ulcer)
* Currently using birth control
* Known allergy to aspirin, non-steroidal anti-inflammatory drugs (NSAIDS) or Sulfa-drugs
* Diabetes
* Cardiac disease or hypertension
* Moderate to severe heartburn (GERD)
* Obesity (BMI greater than 30)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, MD, MPH, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- See also: OHSU Women's Health Research Unit — http://www.ohsuwomenshealth.com/research/index.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects may also have learned about the study from an OHSU Center for Women's Health provider.Visit 1: reviewed of medical history and demographics and vital signs. A blood draw and urine pregnancy test was performed. Eligible subjects returned for the enrollment.
Groups:
- Active Drug Cycle: Group 1: control cycle, placebo cycle, active drug (celecoxib 400 mg orally, daily x1 menstrual cycle) cycle
- Placebo: Group 2: control cycle, celecoxib cycle, placebo cycle orally, daily x1 menstrual cycle
Period: Overall Study
Arm/Group | Active Drug Cycle | Placebo
Started | 7 | 4
Completed | 7 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Drug Cycle | Placebo | Total
Number analyzed (Participants) | 7 | 4 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 27.3 (5.2) | 28.8 (6.1) | 27.85 (0.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Menstrual Cycle Length
Description: Menstrual cycle length was measured by the number of days subjects noted menstruating in their diary entry.
Time Frame: 3 months
Population: Intention to Treat (ITT)
Measure: Mean (Standard Deviation); unit: Days
Groups:
- Active Drug: Active drug(celecoxib 400 mg orally, daily for 1 menstrual cycle) cycle [cycle = length of menstrual cycle]
- Placebo: Placebo cycle orally, daily x1 menstrual cycle [cycle = length of menstrual cycle]
Arm/Group | Active Drug | Placebo
Number analyzed (Participants) | 7 | 4
Days | 28.5 (2.5) | 27.2 (2.4)

ADVERSE EVENTS:
Arm/Group | Active Drug Cycle | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No